CLINICAL TRIAL: NCT00383721
Title: A Randomized, 26-Week, Placebo-Controlled Efficacy and Safety Study With a 26-Week Long-Term Safety Extension, of High- and Medium-Dose Inhaled Mometasone Furoate/Formoterol Fixed-Dose Combination Formulation Compared With Formoterol and High-Dose Inhaled Mometasone Furoate Monotherapy in Subjects With Moderate to Severe COPD
Brief Title: Effects of Mometasone Furoate/Formoterol Combination Versus Formoterol and Mometasone Furoate Alone in Chronic Obstructive Pulmonary Disease (COPD) (Study P04230AM4)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P04230; Doc ID: 3227335,; Eudract No: 2006-002309-30,
Record Dates: First submitted 2006-09-29; First posted 2006-10-03 (Estimated); Results first posted 2011-10-26 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Mometasone Furoate; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MF/F MDI 400/10 mcg BID (Experimental)
  Interventions: Drug: Mometasone furoate/formoterol (MF/F) combination
- MF/F MDI 200/10 mcg BID (Experimental)
  Interventions: Drug: Mometasone furoate/formoterol (MF/F) combination
- MF MDI 400 mcg BID (Experimental)
  Interventions: Drug: Mometasone furoate MDI (MF MDI)
- Formoterol MDI 10 mcg BID (Active Comparator)
  Interventions: Drug: Formoterol MDI
- Placebo MDI BID (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mometasone furoate/formoterol (MF/F) combination — MF/F 400/10 mcg via a metered dose inhaler (MDI) twice daily for 52 weeks
  Other Names: SCH 418131
  Arms: MF/F MDI 400/10 mcg BID
Drug: Mometasone furoate/formoterol (MF/F) combination — MF/F 200/10 mcg via a metered dose inhaler (MDI) twice daily for 52 weeks
  Other Names: SCH 418131
  Arms: MF/F MDI 200/10 mcg BID
Drug: Mometasone furoate MDI (MF MDI) — MF 400 mcg via metered dose inhaler twice daily for 52 weeks
  Other Names: SCH 32088
  Arms: MF MDI 400 mcg BID
Drug: Formoterol MDI — Formoterol 10 mcg via metered dose inhaler twice a day for 52 weeks
  Other Names: Foradil
  Arms: Formoterol MDI 10 mcg BID
Drug: Placebo — Placebo MDI twice a day for 26 weeks
  Arms: Placebo MDI BID

SUMMARY:
This is a randomized, placebo-controlled, parallel-group, multi-site, double-blind study evaluating the efficacy of mometasone furoate/formoterol fumarate (MF/F) metered dose inhaler (MDI) 400/10 mcg twice daily (BID) and MF/F MDI 200/10 mcg BID compared with MF 400 mcg BID and F 10 mcg BID in adults at least 40 years of age, with moderate to severe chronic obstructive pulmonary disease (COPD). All placebo-treated subjects and active-treated subjects who will not participate in the safety extension will be discontinued and will have their Final Visit at Week 26. Subjects who continue into the 26-week safety extension will have their Final Visit at Week 52. Efficacy will be measured by the mean change from Baseline to Week 13 in area under the forced expiratory volume in one second concentration time curve from 0 to 12 hours (FEV1 AUC[0-12hr]) and change from Baseline to Week 13 in AM predose FEV1.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe COPD based on prebronchodilator FEV1/forced vital capacity (FVC) ratio of <=70%.
* At Screening & Baseline, postbronchodilator FEV1 must be >= 60% predicted normal & >=25% predicted normal.
* COPD symptoms for >=24 months.
* >=2 COPD exacerbations requiring course of oral corticosteroid &/or antibiotics within 2-12 months before screening.
* Ex- or current smoker with smoking history >=10 pack years.
* Only albuterol/salbutamol for relief for at least 2 weeks prior to randomization.
* Withdraw from parenteral & oral steroids, anticholinergics, & antibiotics 4 weeks prior to Screening.
* No harm in changing current COPD therapy, willing to discontinue his/her anticholinergics, inhaled corticosteroids (ICS) or ICS/long-acting beta agonists (LABA) at Screening, & transferred to albuterol/salbutamol for relief for 2 weeks prior to Randomization.
* Lab tests conducted at Screening must be acceptable to investigator. Electrocardiogram (ECG) performed at Screening or within 30 days prior to Screening must be acceptable to investigator. Chest X-ray or computerized tomography (CT) scan is acceptable within 12 months prior to Screening must be acceptable to investigator.
* Female of childbearing potential must use birth control. Includes: hormonal contraceptives, intra-uterine device (IUD), condom in combination with spermicide, monogamous relationship with male partner who had vasectomy. Started birth control at least 3 months prior to Screening (exception condom), & must agree to continue. Female who is not currently sexually active must agree/consent to using a method should she become sexually active. Women who have been surgically sterilized or are at least 1 year postmenopausal are not considered to be of childbearing potential. Female must have negative serum pregnancy test at Screening.

Exclusion Criteria:

* Evidence (upon visual inspection) of oropharyngeal candidiasis at Baseline with or without treatment. If there is evidence at Screening, may be treated as appropriate & visit can be scheduled upon resolution. If there is evidence at Baseline, may be treated as appropriate & visit can be rescheduled upon resolution.
* History of renal, hepatic, cardiovascular, metabolic, neurologic, hematologic, ophthalmological, respiratory, gastrointestinal, cerebrovascular, or other which could interfere with study or require treatment which might interfere with study. Examples include (but are not limited to) hypertension treated with beta-blockers), active hepatitis, coronary artery disease, arrhythmia, significant QTc prolongation (ie QTcF or QTcB [Fridericia or Bazett corrections, respectively >500 milliseconds (msecs)]) stroke, severe rheumatoid arthritis, chronic open-angle glaucoma or posterior subcapsular cataracts, acquired immune deficiency syndrome (AIDS), or conditions that may interfere with respiratory function such as asthma, bronchiectasis, cystic fibrosis. Others which are well-controlled & stable (eg hypertension not requiring beta-blockers) will not prohibit participation if appropriate to investigator.
* Allergy/sensitivity to glucocorticosteroids, beta-2 agonists, study drug/excipients.
* Female who is breast-feeding, pregnant, or intends to become pregnant.
* Illicit drug user.
* Human immunodeficiency virus (HIV) positive (testing not conducted).
* Unable to correctly use oral MDI.
* Taking any restricted medications prior to Screening without meeting washout.
* Cannot adhere to permitted concomitant & prohibited medications.
* May not participate in this same study at another investigational site. Cannot participate in different investigational study at any site, during same time.
* Not be randomized into study more than once.
* No person directly associated with administration of study may participate.
* Previously participated in MF/F trial.
* Increase in absolute volume of >=400 milliliters (mL) at Screening or prior to Baseline within 30 minutes after administration of 4 inhalations of albuterol/salbutamol (total dose of 360 to 400 mcg), or nebulized 2.5 mg albuterol/salbutamol.
* Asthma.
* Lobectomy, pneumonectomy or lung volume reduction surgery.
* Lung cancer.
* Requires long-term administration of oxygen (>15 hours/day).
* Alpha-1-antitrypsin deficiency.
* A history and/or presence of intraocular pressure in either eye >=22 millimeters of mercury (mm Hg), glaucoma, and/or posterior subcapsular cataracts. A subject who has undergone incisional or intraocular surgery in which the natural lens is still present in the eye. A subject with a history of penetrating trauma to both eyes. A subject with one or more of the following Lens Opacities Classification System (LOCS) III grades at screening:

  * nuclear opalescence (NO): >=3.0,
  * nuclear color (NC): >=3.0,
  * cortical cataract (C): >=2.0,
  * posterior subcapsular (P): >=0.5.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1196 (Actual)
Dates: Start 2006-09; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maspero J, Cherrez I, Doherty DE, Tashkin DP, Kuna P, Kuo WL, Gates D, Nolte H, Chylack LT Jr. Appraisal of lens opacity with mometasone furoate/formoterol fumarate combination in patients with COPD or asthma. Respir Med. 2014 Sep;108(9):1355-62. doi: 10.1016/j.rmed.2014.04.015. Epub 2014 May 2. PMID 25044280
- [Derived] Tashkin DP, Doherty DE, Kerwin E, Matiz-Bueno CE, Knorr B, Shekar T, Gates D, Staudinger H. Efficacy and safety characteristics of mometasone furoate/formoterol fumarate fixed-dose combination in subjects with moderate to very severe COPD: findings from pooled analysis of two randomized, 52-week placebo-controlled trials. Int J Chron Obstruct Pulmon Dis. 2012;7:73-86. doi: 10.2147/COPD.S29444. Epub 2012 Feb 3. PMID 22334770
- [Derived] Doherty DE, Tashkin DP, Kerwin E, Knorr BA, Shekar T, Banerjee S, Staudinger H. Effects of mometasone furoate/formoterol fumarate fixed-dose combination formulation on chronic obstructive pulmonary disease (COPD): results from a 52-week Phase III trial in subjects with moderate-to-very severe COPD. Int J Chron Obstruct Pulmon Dis. 2012;7:57-71. doi: 10.2147/COPD.S27320. Epub 2012 Feb 3. PMID 22334769

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Week 26, all participants randomized to placebo were to be discontinued, while 75% of participants randomized to an active treatment were randomly selected to participate in the 26-week Treatment Safety Extension. Several placebo-treated participants continued in error into the Treatment Safety Extension.
Groups:
- MF/F MDI 400/10 mcg BID: Mometasone furoate/formoterol fumarate (MF/F) 400/10 mcg via a metered dose inhaler (MDI) twice daily (BID) for 52 weeks.
- MF/F MDI 200/10 mcg BID: MF/F 200/10 mcg via a MDI BID for 52 weeks.
- MF MDI 400 mcg BID: Mometasone furoate (MF) 400 mcg via a MDI BID for 52 weeks.
- F MDI 10 mcg BID: Formoterol fumarate (F) 10 mcg via a MDI BID for 52 weeks.
- Placebo: Placebo MDI BID for 26 weeks.
Period: 26-Week Double-Blind Treatment Period
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo
Started | 225 | 239 | 253 | 243 | 236
Completed | 190 (1 participant listed as "ongoing" since the participant status could not be formally confirmed.) | 202 | 202 | 193 | 169
Not Completed | 35 | 37 | 51 | 50 | 67
Not completed — Adverse Event | 11 | 5 | 7 | 14 | 13
Not completed — Lack of Efficacy | 1 | 3 | 3 | 4 | 8
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1 | 4
Not completed — Participant withdrawal unrelated | 4 | 12 | 15 | 10 | 11
Not completed — Participant withdrawal related | 5 | 3 | 6 | 8 | 9
Not completed — Non-compliance with protocol | 7 | 5 | 4 | 6 | 6
Not completed — Did not meet protocol eligibility | 5 | 6 | 11 | 4 | 13
Not completed — Administrative | 1 | 3 | 3 | 3 | 3
Not completed — Ongoing | 1 | 0 | 0 | 0 | 0
Period: 26-Week Treatment Safety Extension
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo
Started | 145 | 153 | 149 | 148 | 8
Completed | 126 | 136 | 126 | 131 | 8
Not Completed | 19 | 17 | 23 | 17 | 0
Not completed — Adverse Event | 6 | 7 | 10 | 1 | 0
Not completed — Lack of Efficacy | 0 | 2 | 4 | 1 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 1 | 0
Not completed — Participant withdrawal unrelated | 6 | 4 | 2 | 7 | 0
Not completed — Participant withdrawal related | 1 | 1 | 1 | 1 | 0
Not completed — Non-compliance with protocol | 2 | 1 | 1 | 4 | 0
Not completed — Did not meet protocol eligibility | 1 | 0 | 1 | 1 | 0
Not completed — Administrative | 1 | 2 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo | Total
Number analyzed (Participants) | 225 | 239 | 253 | 243 | 236 | 1196
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.1) | 60.1 (9.0) | 60.5 (8.5) | 59.7 (8.7) | 58.8 (9.5) | 59.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 64 | 56 | 61 | 58 | 296
  Male | 168 | 175 | 197 | 182 | 178 | 900

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Time Curve From 0 to 12 Hours (AUC(0-12 Hours)) of Change From Baseline to Week 13 in Forced Expiratory Volume (Liters) in 1 Second (FEV1)
Description: FEV1 AUC was standardized to liters. Endpoint was the last post-baseline non-missing result through Week 13 carried forward.
Time Frame: Baseline to Endpoint (13 weeks)
Population: Intent-to-treat (ITT) population
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo
Number analyzed (Participants) | 216 | 230 | 246 | 236 | 225
Liters
  Baseline | 1.189 (0.408) | 1.195 (0.408) | 1.260 (0.408) | 1.176 (0.408) | 1.205 (0.408)
  Endpoint (Change from Baseline) | 0.179 (0.274) | 0.139 (0.274) | 0.053 (0.274) | 0.092 (0.274) | 0.018 (0.274)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg BID vs MF MDI 400 mcg BID; Test type: Superiority or Other; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg BID vs MF MDI 400 mcg BID; Test type: Superiority or Other; p < 0.001, ANCOVA

2. Primary Outcome: Mean Change From Baseline to Week 13 Endpoint in AM Predose FEV1
Description: Endpoint was the last post-baseline non-missing result through Week 13 carried forward.
Time Frame: Baseline to Endpoint (13 weeks)
Population: ITT population
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo
Number analyzed (Participants) | 215 | 228 | 245 | 235 | 224
Liters
  Baseline | 1.188 (0.408) | 1.194 (0.408) | 1.255 (0.408) | 1.175 (0.408) | 1.205 (0.408)
  Endpoint (Change from Baseline) | 0.098 (0.280) | 0.063 (0.280) | 0.028 (0.280) | 0.049 (0.280) | -0.003 (0.280)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p = 0.062, ANCOVA
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg BID vs F MDI 10 mcg BID; Test type: Superiority or Other; p = 0.583, ANCOVA

3. Secondary Outcome: Change From Baseline to Endpoint in St George's Respiratory Questionaire (SGRQ) Total Score
Description: SGRQ consisted of 76 items aggregated into 3 component scores: symptoms
  (frequency/severity), activity (cause or limited by breathlessness), impact (social functioning, psychological disturbances from airway disease), & total score. Best health scores have a low numeric value. All component scores & total score ranged from 0-100, with a higher score indicating greater disease burden. A 4-point increase over placebo (and Baseline) was considered the minimum clinically important difference. Endpoint was the last post-baseline non-missing result through the 26 week evaluation carried forward.
Time Frame: Baseline to Endpoint (26 weeks)
Population: ITT population
Measure: Least Squares Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo
Number analyzed (Participants) | 211 | 227 | 240 | 231 | 216
Score on a scale
  Baseline | 48.22 (17.49) | 47.29 (17.49) | 48.27 (17.49) | 46.27 (17.49) | 46.59 (17.49)
  Endpoint (Change from Baseline) | -6.04 (13.95) | -7.99 (13.95) | -5.87 (13.95) | -4.93 (13.95) | -2.88 (13.95)
Statistical Analysis 1: Comparison: MF/F MDI 400/10 mcg BID vs Placebo; Test type: Superiority or Other; p = 0.020, ANCOVA
Statistical Analysis 2: Comparison: MF/F MDI 200/10 mcg BID vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Secondary Outcome: Change From Baseline in Proportion of Chronic Obstructive Pulmonary Disease (COPD) Symptom-Free Nights (AM Diary Symptoms)
Description: Prior to the use of study drug rescue medication (in the morning upon awakening) the participant evaluated the COPD symptoms of wheezing, cough, and difficulty breathing. A symptom-free night was defined as a combined score of 0 (no symptoms) across all three COPD symptoms evaluated the following morning. Proportion for Baseline included data from the last week before the first dose. Proportion for Endpoint included data across the entire 26-week treatment period.
Time Frame: Baseline to Endpoint (26 weeks)
Population: ITT population
Measure: Least Squares Mean (Standard Deviation); unit: Proportion of symptom-free nights
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo
Number analyzed (Participants) | 213 | 228 | 242 | 234 | 224
Proportion of symptom-free nights
  Baseline | 0.24 (0.334) | 0.22 (0.334) | 0.24 (0.334) | 0.25 (0.334) | 0.24 (0.334)
  Endpoint (Change from Baseline) | 0.13 (0.29) | 0.17 (0.29) | 0.16 (0.29) | 0.13 (0.29) | 0.12 (0.29)

5. Secondary Outcome: Number of Participants With Partly Stable COPD
Description: Partly stable COPD was a composite measure that included the following COPD
  outcomes: (1) No oral steroid rescue medication; (2) No AM or PM COPD weekly
  average symptom score greater than 2 during at least 7 of 8 weeks; (3) No moderate or severe exacerbations; (4) No unscheduled visits due to COPD worsenings; (5) No study discontinuation due to treatment failure or treatment-related adverse event as determined by the investigator.
Time Frame: Endpoint (26 weeks)
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo
Number analyzed (Participants) | 221 | 235 | 249 | 239 | 232
Participants | 91 | 101 | 92 | 98 | 87

6. Secondary Outcome: Number of Participants With Mild, Moderate, or Severe COPD Exacerbations
Description: Mild = 12 or more inhalations/day of inhaled rescue medication or 2 or more
  nebulized treatments/day of inhaled rescue medication. Moderate = treatment with
  antibiotics or oral steroids. Severe = emergency room treatment or hospitalizations of survival curves. If an event was composed of multiple criteria, the most severe criteria was assigned to the event.
Time Frame: Endpoint (26 weeks)
Population: ITT population
Measure: Number; unit: Participants
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo
Number analyzed (Participants) | 221 | 235 | 249 | 239 | 232
Participants
  Mild | 56 | 53 | 49 | 61 | 64
  Moderate | 24 | 20 | 29 | 33 | 38
  Severe | 3 | 3 | 5 | 2 | 4

ADVERSE EVENTS:
Description: Treatment period for adverse events was 52 weeks for MF/F MDI 400/10 mcg BID,
  MF/F MDI 200/10 mcg BID, MF MDI 400 mcg BID, and F MDI 10 mcg BID and 26
  weeks for placebo.
Arm/Group | MF/F MDI 400/10 mcg BID | MF/F MDI 200/10 mcg BID | MF MDI 400 mcg BID | F MDI 10 mcg BID | Placebo
Serious Adverse Events (participants affected / at risk) | 26/225 | 28/239 | 33/253 | 25/243 | 21/236
Other Adverse Events (participants affected / at risk) | 37/225 | 28/239 | 34/253 | 30/243 | 34/236
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 400/10 mcg BID (N=225) | MF/F MDI 200/10 mcg BID (N=239) | MF MDI 400 mcg BID (N=253) | F MDI 10 mcg BID (N=243) | Placebo (N=236)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cor pulmonale (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cataract subcapsular (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lenticular opacities (Eye disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (2) | 1 (2)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric atrophic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amoebic dysentery (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (6) | 1 (1) | 4 (5) | 4 (5) | 1 (1)
Pumonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal abcess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Collapse of lung (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 8 (10) | 12 (14) | 9 (10) | 13 (14)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF/F MDI 400/10 mcg BID (N=225) | MF/F MDI 200/10 mcg BID (N=239) | MF MDI 400 mcg BID (N=253) | F MDI 10 mcg BID (N=243) | Placebo (N=236)
Nasopharyngitis (Infections and infestations) | 13 (16) | 9 (11) | 14 (21) | 12 (13) | 9 (11)
Upper respiratory tract infection (Infections and infestations) | 18 (20) | 8 (12) | 8 (10) | 10 (13) | 11 (13)
Headache (Nervous system disorders) | 9 (16) | 12 (24) | 16 (21) | 11 (29) | 14 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to publish or publicly present results. The investigator agrees not to publish or publicly present any interim results without prior written consent of the sponsor. The investigator agrees to provide to the sponsor 45 days before submission for publication that

report results of the study. The sponsor shall have the right to review & comment with respect to publications, abstracts, slides, & manuscripts & the right to review & comment on the data & presentation.